CLINICAL TRIAL: NCT05862792
Title: Impact of Liposomal Bupivacaine on Post-operative Pain, Opioid Use, and Swallow Function in Transoral Robotic Surgery
Brief Title: Liposomal Bupivacaine and Transoral Robotic Surgery
Status: Recruiting | Type: Observational
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-0739
Record Dates: First submitted 2023-01-09; First posted 2023-05-17 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Oropharyngeal Cancer; Dysphagia, Oropharyngeal; Post Operative Pain; Transoral Robotic Surgery
Keywords: oropharyngeal cancer; squamous cell carcinoma; postoperative pain; transoral robotic surgery
MeSH Terms: conditions — Oropharyngeal Neoplasms; Deglutition Disorders; Pain, Postoperative; Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- TORS + Liposomal Bupivacaine + Postoperative Antipyretics and Opioids Group: Per standard of care, at the conclusion of the TORS procedure, liposomal bupivacaine will be injected into the surgical bed- (bupivacaine liposome suspension 1.3% [13.3 mg/mL], intramuscular) in this group. Possible injection sites include the base of tongue and/or tonsil. Total dose injected will be 3-4 mL. Subjects will also be given a pain regimen including:
  1. Tylenol 650 mg every 4 hours as needed for mild pain
  2. Oxycodone 5 mg every 4 hours as needed for moderate pain
  3. Morphine 2mg every 3 hours as needed for breakthrough pain
  The treatment type (TORS +/- Liposomal Bupivacaine + Postoperative Antipyretics and Opioids) is determined by the subject's surgeon based on his standard practice.
  Interventions: Drug: Liposomal bupivacaine
- TORS + Postoperative Antipyretics and Opioids Group: Per standard of care, subjects in this group will only be given a pain regimen including:
  1. Tylenol 650 mg every 4 hours as needed for mild pain
  2. Oxycodone 5 mg every 4 hours as needed for moderate pain
  3. Morphine 2mg every 3 hours as needed for breakthrough pain
  The treatment type (TORS +/- Liposomal Bupivacaine + Postoperative Antipyretics and Opioids) is determined by the subject's surgeon based on his standard practice.

INTERVENTIONS:
Drug: Liposomal bupivacaine — We will inject liposomal bupivacaine into the surgical bed.
  Other Names: EXPAREL
  Groups: TORS + Liposomal Bupivacaine + Postoperative Antipyretics and Opioids Group

SUMMARY:
This study is for patients with oropharyngeal squamous cell carcinoma. We want to learn more about how we can optimize pain control in patients who undergo transoral robotic surgery (TORS) for oropharyngeal squamous cell carcinoma. Our goal is to determine if a local anesthetic called EXPAREL® (Liposomal Bupivacaine) impacts postsurgical pain and swallow function in patients with oropharyngeal squamous cell carcinoma undergoing TORS. EXPAREL® is an FDA-approved anesthetic drug that provides long-lasting and precise pain relief when injected into the surgical wound. Our study team wants to determine if injecting EXPAREL® into the surgical wound will provide better pain relief and swallow function when compared to patients who do not undergo postoperative EXPAREL® injection. Both options for postoperative pain control are considered standard of care for patients undergoing TORS.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, greater than or equal to 18 years of age; Patients of all genders; Patients undergoing transoral robotic surgery; Patient who are able and willing to give consent

Exclusion Criteria:

* Patients with an allergy to Bupivacaine or other amide anesthetics; Patients with a carnitine deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing TORS
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Control | 3 months
  We will be measuring subjects' postoperative maximum visual analog pain scores on each postoperative day.
  Scale: 0-10, 0 represents no pain and 10 represents the worst pain
Postoperative Dysphagia with Endoscopic Swallow Study | 3 months
  Patients will undergo a functional endoscopic swallow study with a speech language pathologist during their first postoperative visit.
Postoperative Dysphagia with Dysphagia Survey | 3 months
  Patients will undergo an evaluation of their swallow function via the MD Anderson Dysphagia Inventory survey with a speech language pathologist during their first postoperative visit.

SECONDARY OUTCOMES:
Postoperative Pain Medication Usage | 3 months
  We will be measuring the doses of pain medication that patients requiring during their postoperative course.

CONTACTS AND LOCATIONS:
Locations (1):
- Geisinger Medical Center, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No